CLINICAL TRIAL: NCT03919318
Title: Effect of Two Different Calcium Silicate Based and One Epoxy Resin-based Root Canal Sealers on Postoperative Pain After Root Canal Treatments
Brief Title: Postoperative Pain After the Use of Different Root Canal Sealers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Tuğrul Aslan, Assisstant Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/08
Record Dates: First submitted 2019-04-14; First posted 2019-04-18 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; Endoseal MTA; Endosequence BC; AH Plus; Root canal filling; endodontic treatment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AH-Plus (Experimental)
  Interventions: Other: Root Canal Filling Sealers
- EndoSeal MTA (Experimental)
  Interventions: Other: Root Canal Filling Sealers
- Endosequence BC Sealer (Experimental)
  Interventions: Other: Root Canal Filling Sealers

INTERVENTIONS:
Other: Root Canal Filling Sealers — Root Canal Obturation

SUMMARY:
This study evaluated the postoperative pain after the endodontic treatment using AH Plus, Endoseal MTA and EndoSequence BC sealers in root canal obturation.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 - 60 years of age,
* Good oral hygiene,
* Have not taken any analgesics in the last day,
* Have not taken antibiotics in the last week,
* Patients diagnosed with asymptomatic irreversible pulpitis caused by deep carious lesion on the mandibular first or second molar teeth.
* A prolonged positive response to cold vitality tests,
* The presence of pulp, which is exposed during caries removing and bleeding with a dense and thick consistency.
* The periapical region was healthy in radiographic diagnosis.

Exclusion Criteria:

* Devital teeth that have no response to pulp test,
* The presence of advanced periodontal disease,
* Having a systemic disease that requires antibiotic prophylaxis,
* Radiographically more than 30° root inclination, presence of clear apex, presence of calcification, presence of root resorption,
* The need for root canal treatment which is mesial and/or distal neighbour of the tooth to be treated,
* The presence of a sinus tract in the relevant tooth region,
* Having systemic diseases that reduce immune system resistance,
* Participants with allergic sensitivity to materials and agents that should be used during the root canal treatment,
* Allergic sensitivity to local anesthetics,
* Pregnant participants or participants in the lactation period,
* Over preparation or over filling during treatment,
* Teeth which cannot be applied a rubber-dam,
* Teeth which was damaged enough to require coronal fiber post application,
* Sensitive to Ibuprofen based analgesics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 6th hours. | 6th hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 12th hours. | 12th hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 24th hours. | 24th hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 48th hours. | 48th hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 3rd days. | 3rd days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 4th days. | 4th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 5th days. | 5th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 6th days. | 6th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different endodontic sealers: VAS (Visual Analogue Scale) at 7th days. | 7th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.

SECONDARY OUTCOMES:
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 6th hours. | 6th hours
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 12th hours. | 12th hours
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 24th hours. | 24th hours
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 48th hours. | 48th hours
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 3rd days. | 3rd days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 4th days. | 4th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 5th days. | 5th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 6th days. | 6th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different endodontic sealers at 7th days. | 7th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"

CONTACTS AND LOCATIONS:
Overall Officials: Tuğrul Aslan, PHD. Dr., Study Director — Erciyes University, Faculty of Dentistry
Locations (1):
- Erciyes University, Faculty of Dentistry, Kayseri, İç Anadolu, Turkey (Türkiye)

REFERENCES:
- [Background] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915
- [Background] Atav Ates A, Dumani A, Yoldas O, Unal I. Post-obturation pain following the use of carrier-based system with AH Plus or iRoot SP sealers: a randomized controlled clinical trial. Clin Oral Investig. 2019 Jul;23(7):3053-3061. doi: 10.1007/s00784-018-2721-6. Epub 2018 Nov 5. PMID 30397735